CLINICAL TRIAL: NCT04760600
Title: Role of Parasitic Infection in Inflammatory Bowel Disease and Irritable Bowel Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, marina gamil shwqi, principle investigator, Assiut University
Other Study IDs: role of parasites in ibd ibs
Record Dates: First submitted 2021-02-05; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-01

CONDITIONS: Parasite IBS IBD

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- IBD GROUPS: PATIENT WITH IBD DISEASE
- IBS GROUP: PATIENT WIT IBS DISEASE
- CONTROL 1: CONTROL WITH POSITIVE PARASITIC INFECTION AN POSITIVE GIT SYMTOMS
- CONTROL2: HEALTHY VOLUNTEARS

SUMMARY:
Role of parasitic infection in Inflammatory bowel disease and Irritable bowel The burden of the parasitic disease is in-direct relation with the health and nutritional status of the host, inducing not only parasite-specific immunity but also can modify the host's immune responses . Many parasites can imitate inflammatory bowel disorders and some studies showed that infection with parasites can improve disorders like IBD or moderate the symptoms of inflammatory bowel disorders . Even though, many studies have shown that gastrointestinal infection is an important risk factor for the development of IBS

DETAILED DESCRIPTION:
1. Detect the prevalence of parasite/s associated with Inflammatory bowel diseases (IBD) and Irritable bowel syndrome (IBS) in comparison with control subjects.
2. Evaluating the effect of the parasite on the course and prognosis of the diseases.
3. Evaluating the effect of the antiparasitic drugs on the course and prognosis of the diseases.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IBD will be confirmed using

  1. standard clinical,
  2. endoscopic,
  3. radiographic and4 pathological criteria according to the Montreal classification of the extent and severity of IBD
* Diagnosis of IBS will depend on Rome IV criteria

  1. Recurrent abdominal pain on average at least 1 day/week in the last 3 months,
  2. associated with two or more of the following criteria:
  3. Related to defecation;
  4. Associated with a change in the frequency of stool and/ or Associated with a change in the form (appearance) of stool.

Exclusion Criteria:

* any patient who received antipiotic or antiparasitic drug within the past 4 weeks

Ages: 17 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Diagnosis of IBD will be confirmed using standard clinical, endoscopic, radiographic and pathological criteria according to the Montreal classification of the extent and severity of IBD The activity of the disease will be measured using the Mayo Clinic score consisting of 4 items: stool frequency, rectal bleeding, findings of flexible proctosigmoidoscopy, and patient's functional assessment Diagnosis of IBS will depend on Rome IV criteria Recurrent abdominal pain on average at least 1 day/week in the last 3 months, associated with two or more of the following criteria: Related to defecation; Associated with a change in the frequency of stool and/ or Associated with a change in the form (appearance) of stool.
  * any patient who received antipiotic or antiparasitic drug within the past 4 weeks not taken
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Detect the prevalence of parasite/s associated with Inflammatory bowel diseases (IBD) and Irritable bowel syndrome (IBS) in comparison with control subjects. | baseline
  Detect the prevalence of parasite/s associated with Inflammatory bowel diseases (IBD) and Irritable bowel syndrome (IBS) in comparison with control subjects.by making stool analysis and clinical examination

SECONDARY OUTCOMES:
measure the effect of the antiparasitic drugs on the course and prognosis of the diseases | baseline
  giving the patient antiparasitic drug and measure the effect of anti parasitic drug on course and prognosis of disease

CONTACTS AND LOCATIONS:
Overall Officials: rasha hassan, Principal Investigator — Assiut University; mona mostafa, Principal Investigator — Assiut University
Locations (1):
- Marina Gamil Shwqi, Asyut, Egypt

REFERENCES:
- See also: Human Intestinal Parasites — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC2754014/
- See also: Comparative pathobiology of the intestinal protozoan parasites giardia lamblia, entamoeba histolytica, and cryptosporidium parvum — http://www.mendeley.com/catalogue/7d32c086-0fd2-3c70-a8f6-456b2737bdaa/?utm_source=desktop&utm_medium=1.19.4&utm_campaign=open_catalog&userDocumentId=%7Bce3e00ed-dfc4-436d-98ea-beb2dd8f2961%7D
- See also: Opportunistic infections due to inflammatory bowel disease therapy — http://www.mendeley.com/catalogue/751a62fa-7a37-31b6-85ec-176f042b5e4d/?utm_source=desktop&utm_medium=1.19.4&utm_campaign=open_catalog&userDocumentId=%7B7ea29a48-e517-4237-9dc4-b0d319284902%7D
- See also: Prevalence of Intestinal Parasitic Infections among the Bulgarian Population Over a Three Year Period — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC6996262/
- See also: Soil-transmitted helminth infections: updating the global picture — http://pubmed.ncbi.nlm.nih.gov/14642761/
- See also: Chronic intestinal inflammation: inflammatory bowel disease and colitis-associated colon cancer — https://pubmed.ncbi.nlm.nih.gov/22586430/
- See also: Clinical and Mechanistic Characteristics of Current JAK Inhibitors in IBD — http://pubmed.ncbi.nlm.nih.gov/33295611/